CLINICAL TRIAL: NCT06961279
Title: Resveratrol Stimulates Insulin Sensitivity, and Changes Microbiota Taxonomy and Serum Metabolomics in Participants With Obesity and Insulin Resistance
Brief Title: Resveratrol Stimulates Insulin Sensitivity in Subjects With Obesity and Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1099A
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resveratrol (Experimental): Resveratrol capsules of 75 mg each, 150 mg/day
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): Maltodextrin capsules, administered orally once every 12 hours
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol — Administered orally once every 12 hours
  Arms: Resveratrol
Dietary Supplement: Placebo — Administered orally once every 12 hours
  Arms: Placebo

SUMMARY:
There is evidence that resveratrol can improve insulin resistance in rodents and humans with obesity and it can also improve muscle mitochondrial content mediated through activation of AMPK. However, little is known if this improvement is associated with changes in the gut microbiota and how gut microbiota is associated with serum metabolites after consumption of resveratrol. In the present study, the investigators show that the consumption of resveratrol for 2 months could influence insulin sensitivity in subjects with obesity. This effect will be accompanied by a modification of the microbiota taxonomy and the metabolites derived from this. Consequently, there will be a reduction in metabolic endotoxemia accompanied by an increase in AMP-activated protein kinase (AMPK) phosphorylation and the expression of genes of mitochondrial biogenesis in skeletal muscle.

DETAILED DESCRIPTION:
The investigators included 38 participants who met the following inclusion criteria: adults between 20 and 60 years of age with a diagnosis of HOMA-IR index greater than 2.5, and BMI ≥30 and ≤ 40 kg / m2 and who signed the consent letter. Participants who had any added pathology, pregnancy, smoking or consumed medications were excluded. Once the letter of informed consent was accepted, the patients were assigned to the respective treatment group. These individuals were advised to consume the recommended diet for subjects with obesity. Participants were randomly distributed to consume a) placebo treatment or b) resveratrol capsules (150 mg/day). The participants were followed for 2 months. In the pre-randomization visit, informed consent letters were given, and blood samples were taken to evaluate glucose concentration, lipid profile and serum insulin, blood pressure, body weight and height and body composition. The presence of insulin resistance was determined by means of the HOMA-IR index. For the first visit body composition, other biochemical parameters such as protein c reactive, alanine transaminase, aspartate transaminase, hemoglobin glycosylated, hormones as leptin and adiponectin, free fatty acids in serum, malondialdehyde in serum, lipopolysaccharide in serum, short chain fatty acids in feces, fecal microbiota and serum metabolomics were determined. After 2 months, the same variables were assessed, and an expert surgeon in the operating room performed a vastus lateralis muscle biopsy, then protein extraction was performed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female.
* Between 20 and 60 years
* BMI ≥ 30 and ≤ 40 kg/m2
* Presence of insulin resistance (HOMA-IR index ≥ 2.5)
* Willing and able to sign written informed consent prior to trial entry

Exclusion Criteria:

* Patients with any type of diabetes.
* Patients with kidney disease diagnosed by a medical or with creatinine> 1.3 mg / dL for men and > 1.1 mg / dL for women and / or BUN> 20 mg / dL.
* Patients with acquired diseases that produce obesity and diabetes secondarily.
* Patients who have suffered a cardiovascular event.
* Patients with gastrointestinal diseases.
* Weight loss > 3 kg in the last 3 months.
* Catabolic diseases such as cancer and acquired immunodeficiency syndrome.
* Pregnancy status.
* Antibiotic consumption 3 months prior to the study.
* Be an undergraduate or graduate student within the Institute.
* Positive smoking.
* Drug treatment:

  * Antihypertensive drugs or treatment
  * Treatment with hypoglycemic agents or insulin and antidiabetic drugs.
  * Treatment with statins, fibrates or other drugs to control dyslipidemia.
  * Use of antibiotics in the three months prior to the study.
  * Use of steroid drugs, chemotherapy, immunosuppressants, or radiation therapy.
  * Anorexigenic or that accelerate weight loss such as sibutramine or orlistat.
  * Probiotic, prebiotic or symbiotic supplements.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-09-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Baseline to 2 months
  Measurement of insulin by an oral glucose tolerance test.

SECONDARY OUTCOMES:
Fecal microbiota | Baseline to 2 months
  Composition, abundance and diversity of fecal microbiota by sequencing 16s rRNA gene
Glucose metabolism profile | Baseline to 2 months
  Serum glucose (mg/dL)
Insulin (µUI/ml) | Baseline to 2 months
  Serum insulin
Triglycerides | Baseline to 2 months
  serum triglycerides (mg/dL)
Total cholesterol | Baseline to 2 months
  serum total cholesterol (mg/dL)
LDL cholesterol | Baseline to 2 months
  serum LDL cholesterol (mg/dL)
HDL cholesterol | Baseline to 2 months
  serum HDL cholesterol (mg/dL)
Antioxidant profile | Baseline to 2 months
  Serum malondialdehyde (MDA) (nmol/mL)
Body weight | Baseline to 2 months
  body wight (kg)
Blood pressure | Baseline to 2 months
  blood pressure (mmHg)
Change in PGC1α content | Through study completion, an average of 2 months
  Measure of PGC1α protein content in skeletal muscle tissue taken by biopsy
Change in AMPK content | Through study completion, an average of 2 months
  Measure of AMPK protein content in skeletal muscle tissue taken by biopsy
Succinate dehydrogenase | Through study completion, an average of 2 months
  Fold change in succinate dehydrogenase activity in skeletal muscle tissue taken by biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Armando R Tovar, Dr., Principal Investigator — INCMNSZ
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No